CLINICAL TRIAL: NCT04995120
Title: Induction Chemotherapy and Toripalimab Followed by Surgery or Radiotherapy for Larynx Preservation in Resectable Laryngeal/Hypopharyngeal Carcinoma
Brief Title: Induction Chemotherapy and Toripalimab for Larynx Preservation in Resectable Laryngeal/Hypopharyngeal Carcinoma
Acronym: INSIGHT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiayun He, MD, M.D., professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Larynx-IO 1.0; 2103232-1 (Other: IRB of Fudan Univeristy Shanghai Cancer Center)
Record Dates: First submitted 2021-07-25; First posted 2021-08-06 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Laryngeal Cancer; Hypopharynx Cancer; Laryngeal Neoplasms
Keywords: Induction chemotherapy; Checkpoint inhibitor; PD-1 inhibitor; Toripalimab; Larynx preservation
MeSH Terms: conditions — Laryngeal Neoplasms; Hypopharyngeal Neoplasms | interventions — toripalimab; 130-nm albumin-bound paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Induction chemotherapy and Toripalimab (Experimental): Induction chemotherapy TP regimen combined with Toripalimab for 3 cycles: Toripalimab 240mg d1, Paclitaxel 175mg/m2 d2 or Nab-Paclitaxel 260mg/m2 d2，Cisplatin 25mg/m2 d2-4 q3w.
  Response rate of primary tumor is evaluated using laryngoscopy and head and neck MRI after 3 cycles of induction therapy. If ORR of primary tumor is CR/PR, then chemoradiation is conducted, followed by maintenance therapy of Toripalimab for 8 cycles (6 months). Otherwise, surgery is conducted (laryngeal preservation surgery is preferred), followed by adjuvant radiation/chemoradiation and then maintenance therapy of Toripalimab for 8 cycles.
  Interventions: Drug: chemotherapy TP regimen combined with Toripalimab

INTERVENTIONS:
Drug: chemotherapy TP regimen combined with Toripalimab — Induction chemotherapy TP regimen combined with Toripalimab for 3 cycles: Toripalimab 240mg d1, Paclitaxel 175mg/m2 d2 or Nab-Paclitaxel 260mg/m2 d2，Cisplatin 25mg/m2 d2-4 q3w.
  Response rate of primary tumor is evaluated using laryngoscopy and head and neck MRI after 3 cycles of induction therapy. If overall response rate of primary tumor is complete response or partial response, then chemoradiation is conducted, followed by maintenance therapy of Toripalimab for 8 cycles (6 months). Otherwise, surgery is conducted (laryngeal preservation surgery is preferred), followed by adjuvant radiation/chemoradiation and then maintenance therapy of Toripalimab for 8 cycles.
  Other Names: Paclitaxel or Nab-Paclitaxel; Cisplatin

SUMMARY:
The aim of this study is to define whether combination of induction chemotherapy and PD-1 inhibitor (Toripalimab) improve the rate of larynx preservation, for patients with resectable laryngeal/hypopharyngeal carcinoma.

DETAILED DESCRIPTION:
Historically, induction chemotherapy could provide a chance of larynx preservation for approximate 60-70% of patients with locally advanced laryngeal/hypopharyngeal carcinoma. Recently, phase I-II clinical studies demonstrated excellent pathological response of induction PD-1 inhibitor with/without chemotherapy for locally advanced head and neck cancer. The aim of this study is to define whether combination of induction chemotherapy and PD-1 inhibitor (Toripalimab) improve the rate of larynx preservation, for patients with resectable laryngeal/hypopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, resectable locally advanced laryngeal/hypopharyngeal squamous cell carcinoma (T2-4a, N0-resectable N3, M0);
* Age between 18-75 years;
* Signed inform consent;
* Had at least one measurable lesion according to RECIST 1.1 criteria
* Anticipated overall survival more than 3 months;
* Satisfactory performance status: ECOG (Eastern Cooperative Oncology Group) scale 0-1;
* Normal organ function;
* HBV DNA<500 IU/mL（or 2500 copies/mL）and HCV RNA negative ;
* Male and no pregnant female, able to adapt birth control methods during treatment.

Exclusion Criteria:

* Hypersensitivity to Toripalimab, Paclitaxel, Nab-Paclitaxel and Cisplatin;
* Suffered from malignant tumors, except cervical carcinoma in situ, papillary thyroid carcinoma, or skin cancer (non- melanoma) within five years;
* Severe, uncontrolled heart disease;
* Receive vaccine or live vaccine within 28 days prior to signing the informed consent;
* Equivalent dose more than prednisone 10mg/d or other immunosuppressive treatments within 28 days prior to signing the informed consent;
* Surgery or trauma within 28 days prior to signing the informed consent;
* Received other immune checkpoint inhibitors previously;
* Severe, uncontrolled infections within 28 days of prior to signing the informed consent;
* Active, known or suspected autoimmune disease; Type I Diabetes, hypothyroidism those only need hormone replacement therapy, vitiligo or inactive asthma who don't need systemic therapy can recruit;
* History of interstitial lung disease;
* HIV positive;
* Hepatitis B surface antigen (HBsAg) positive and HBV-DNA ≥500IU/ml, or 2500cps/ml; Positive HCV RNA;
* Other diseases which may influence the safety or compliance of the clinical trial, such as mental illness, or their family and society factors;
* Women of child-bearing potential who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Laryngeal Preservation rate at 3-month post-radiotherapy | 3-month post-radiotherapy
  defined as the absence of any residual disease that would justify salvage total laryngectomy

SECONDARY OUTCOMES:
Overall response rate of induction therapy | 2 weeks after the 3th cycle of induction therapy
  Overall response rate of induction therapy evaluated by head and neck MR/CT, laryngoscopy using Recist 1.1 Criteria
Overall response rate of treatment | 3 months post-radiotherapy
  Overall response rate of treatment evaluated by head and neck MR/CT, laryngoscopy using Recist 1.1 Criteria
Pathological complete response rate of the patients receiving surgical resection | Within 3 weeks after surgery
  Pathological complete response rate of the patients receiving surgical resection, evaluated by experienced pathologists
Major pathologic response rate of the patients receiving surgical resection | Within 3 weeks after surgery
  Major pathologic response rate, defined as no more than 10% of residual viable tumor, evaluated by experienced pathologists.
Overall survival rate at 1 year | One year post-radiotherapy
  Overall survival rate at 1 year
Overall survival rate at 2 year | Two year post-radiotherapy
  Overall survival rate at 2 year
Progression-free survival rate at 1 year | One year post-radiotherapy
  Progression-free survival rate at 1 year
Progression-free survival rate at 2 year | Two year post-radiotherapy
  Progression-free survival rate at 2 year
Laryngeal Preservation rate at 1 year | One year post-radiotherapy
  Laryngeal Preservation rate at 1 year
Laryngeal Preservation rate at 2 year | Two year post-radiotherapy
  Laryngeal Preservation rate at 2 year
Adverse Effect | One year post-radiotherapy
  Adverse Effect, evaluated by CTCAE 4.0.03

OTHER OUTCOMES:
Laryngeal Preservation rate at 3 month post-radiotherapy by different biomarker subgroups | 3-month post-radiotherapy
  Experimental Biomarker Analysis: the relationship with different biomarkers and 3 month laryngeal preservation rate
Overall response rate of induction therapy, by different biomarker subgroups | 2 weeks after the 3th cycle of induction therapy
  Experimental Biomarker Analysis: the relationship with different biomarkers and overall response rate of induction therapy
Pathological complete response rate by different biomarker subgroups | Within 3 weeks after surgery
  Experimental Biomarker Analysis: the relationship with different biomarkers and pathological complete response rate of the patients receiving surgical resection
Major pathologic response rate by different biomarker subgroups | Within 3 weeks after surgery
  Experimental Biomarker Analysis: the relationship with different biomarkers and major pathologic response rate of the patients receiving surgical resection

CONTACTS AND LOCATIONS:
Overall Officials: Xiayun He, M.D., Principal Investigator — Fudan Universtiy Shanghai Cancer Center; Yu Wang, M.D., Principal Investigator — Fudan Universtiy Shanghai Cancer Center
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janoray G, Pointreau Y, Garaud P, Chapet S, Alfonsi M, Sire C, Jadaud E, Calais G. Long-term Results of a Multicenter Randomized Phase III Trial of Induction Chemotherapy With Cisplatin, 5-fluorouracil, +/- Docetaxel for Larynx Preservation. J Natl Cancer Inst. 2015 Dec 16;108(4):djv368. doi: 10.1093/jnci/djv368. Print 2016 Apr. PMID 26681800
- [Background] Department of Veterans Affairs Laryngeal Cancer Study Group; Wolf GT, Fisher SG, Hong WK, Hillman R, Spaulding M, Laramore GE, Endicott JW, McClatchey K, Henderson WG. Induction chemotherapy plus radiation compared with surgery plus radiation in patients with advanced laryngeal cancer. N Engl J Med. 1991 Jun 13;324(24):1685-90. doi: 10.1056/NEJM199106133242402. PMID 2034244
- [Background] Forastiere AA, Zhang Q, Weber RS, Maor MH, Goepfert H, Pajak TF, Morrison W, Glisson B, Trotti A, Ridge JA, Thorstad W, Wagner H, Ensley JF, Cooper JS. Long-term results of RTOG 91-11: a comparison of three nonsurgical treatment strategies to preserve the larynx in patients with locally advanced larynx cancer. J Clin Oncol. 2013 Mar 1;31(7):845-52. doi: 10.1200/JCO.2012.43.6097. Epub 2012 Nov 26. PMID 23182993
- [Background] Lefebvre JL, Pointreau Y, Rolland F, Alfonsi M, Baudoux A, Sire C, de Raucourt D, Malard O, Degardin M, Tuchais C, Blot E, Rives M, Reyt E, Tourani JM, Geoffrois L, Peyrade F, Guichard F, Chevalier D, Babin E, Lang P, Janot F, Calais G, Garaud P, Bardet E. Induction chemotherapy followed by either chemoradiotherapy or bioradiotherapy for larynx preservation: the TREMPLIN randomized phase II study. J Clin Oncol. 2013 Mar 1;31(7):853-9. doi: 10.1200/JCO.2012.42.3988. Epub 2013 Jan 22. PMID 23341517
- [Background] Weiss J, Gilbert J, Deal AM, Weissler M, Hilliard C, Chera B, Murphy B, Hackman T, Liao JJ, Grilley Olson J, Hayes DN. Induction chemotherapy with carboplatin, nab-paclitaxel and cetuximab for at least N2b nodal status or surgically unresectable squamous cell carcinoma of the head and neck. Oral Oncol. 2018 Sep;84:46-51. doi: 10.1016/j.oraloncology.2018.06.028. Epub 2018 Jul 19. PMID 30115475